CLINICAL TRIAL: NCT05382403
Title: Novel Vacuum-Induced Hemorrhage Control for Postpartum Hemorrhage: a Multicenter Randomized Trial
Brief Title: Novel Vacuum-Induced Hemorrhage Control for Postpartum Hemorrhage
Acronym: NOVIC
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Women and Infants Hospital of Rhode Island (Other)
Collaborators: Washington University School of Medicine (Other); University of Ghana (Other); Kwame Nkrumah University of Science and Technology (Other)
Responsible Party: Principal Investigator, Methodius Tuuli, Professor and Chair of Obstetrics and Gynecology, Women and Infants Hospital of Rhode Island
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PACTR202204852865149
Record Dates: First submitted 2022-05-15; First posted 2022-05-19 (Actual); Last update posted 2023-12-21 (Actual); Status verified 2023-12

CONDITIONS: Postpartum Hemorrhage; Maternal Death
MeSH Terms: conditions — Postpartum Hemorrhage; Maternal Death | interventions — Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Jada® System (Experimental): Patients in this group will have the Jada® System applied when the initial medical treatment fails, and estimated blood loss reaches 1000 mL. It is a U.S. FDA-cleared device intended for treatment of PPH when conservative management is warranted.
  Interventions: Device: Jada® System
- Standard care (Active Comparator): Patients in this group will receive care according to the treatment algorithm for PPH from uterine atony at the two teaching hospitals in Ghana. Possible interventions include additional uterotonics, tranexamic acid, and condom catheter balloon uterine tamponade. If bleeding is uncontrolled, patients will have surgical intervention with options of uterine vascular ligation, uterine compression sutures or hysterectomy
  Interventions: Other: Standard care

INTERVENTIONS:
Device: Jada® System — This is a U.S. FDA-cleared device intended for treatment of PPH when conservative management is warranted. The device is made of medical grade silicone. The distal end, which is placed in the uterus, is an elliptical loop. The circular cervical seal, just outside the external cervical os, is filled with 60 - 120 mL sterile water. Low-level vacuum (80 ± 10 mm Hg) is applied and pooled blood is evacuated from the uterus as it collapses. Once there is no bleeding, the device remains in the uterus for at least 1 hour. The suction is then disconnected, the seal emptied of water, the device left in place, and the patient monitored for an additional 30 minutes. If bleeding remains controlled, the device is removed. If bleeding is uncontrolled with the Jada® System patients will have surgical intervention with options of uterine vascular ligation, uterine compression sutures or hysterectomy.
  Arms: Jada® System
Other: Standard care — Patients in this group will receive care according to the treatment algorithm for PPH from uterine atony at the two teaching hospitals in Ghana. Possible interventions include additional uterotonics, tranexamic acid, and condom catheter balloon uterine tamponade. If bleeding is uncontrolled, patients will have surgical intervention with options of uterine vascular ligation, uterine compression sutures or hysterectomy.
  Arms: Standard care

SUMMARY:
This will be the first, definitive, randomized control trial (N=424) to test the hypothesis that the Jada® System is effective, safe and cost-effective in treating PPH, compared to standard care.

DETAILED DESCRIPTION:
Every year, 130 million women deliver babies around the world, and an estimated 14 million (11%) experience postpartum hemorrhage (PPH), recently redefined as a cumulative blood loss of 1000 ml or more or blood loss associated with signs or symptoms of hypovolemia, irrespective of the route of delivery. PPH is the leading cause of maternal mortality worldwide, responsible for 25% of maternal deaths from obstetric causes, with 99% occurring in low and middle income countries (LMICs). Although PPH has multiple causes, the most common is uterine atony when the uterus fails to adequately contract after childbirth, accounting for 70% of all PPH. Active management of the third stage of labor, consisting of administering prophylactic uterotonics, controlled cord traction, and uterine massage after delivery, reduces the incidence of PPH by approximately 66%. These conservative measures facilitate the normal postpartum tetanic myometrial contractions that constrict the placental bed vasculature. When PPH occurs in spite of these preventive measures, therapeutic options include additional uterotonics (medical), uterine tamponade (mechanical) and surgical interventions (vascular ligation, uterine compression sutures and hysterectomy).

Uterine balloon tamponade is often the second line therapy when medical management is unsuccessful and is achieved with inflatable devices inserted into the uterus to exert outward compression on the uterine walls. Despite its widespread use, its mechanism is counterintuitive to the physiologic uterine contraction that occurs after delivery to control bleeding. Its use is further limited by prolonged treatment times (typically 12-24 hours), urinary tract occlusion, and inability to reveal any continuing bleeding. Low-cost options most commonly condom catheters are used in LMICs, but two recent randomized trials showed no improvement in maternal outcomes and possible harm. Thus, there is an urgent need for effective and safe treatment options to reduce the burden of PPH particularly in LMICs.

The Jada® System (Alydia Health, Menlo Park, CA, USA) is a novel U.S. FDA-cleared intrauterine vacuum-induced hemorrhage-control device specifically designed for rapid treatment of PPH. It mimics postpartum physiology by applying low-level intrauterine negative pressure to facilitate uterine compressive forces for constriction of blood vessels to achieve hemostasis. Preliminary data from two studies have shown promising results. The device was first evaluated in a feasibility case series (n=10) in Indonesia and showed rapid treatment of abnormal postpartum uterine bleeding.6 The second larger study, a multicenter single-arm trial (n=106) in the United States, confirmed quick and definitive control of bleeding in 94% of cases within a median time of 3 minutes and few adverse events. While promising, these data are limited by lack of control groups, possible selection bias and the modest sample sizes which preclude definitive conclusions regarding the relative effectiveness and safety of the Jada® System.

We propose the first, definitive, randomized control trial (N=424) to test the hypothesis that the Jada® System is effective, safe and cost-effective in treating PPH, compared to standard care. A multidisciplinary team of investigators with expertise in obstetrics, global health and clinical trials will enroll 424 women in two high volume obstetric units in Ghana, a LMIC with high PPH burden, to pursue the following specific aims:

Primary Aim: Evaluate the effectiveness of the Jada® System, compared to standard care, in treating PPH.

Secondary Aim 1: Assess the safety of the Jada® System, compared to standard care, in treating PPH.

Secondary Aim 2: Estimate the cost-effectiveness of the Jada® System, compared to standard care, in treating PPH.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older
* Delivery at 34 weeks or greater
* Cumulative blood loss >1000ml within 24 hours after delivery
* Uterine atony
* Receipt of first-line uterotonics
* Cervix at least 3cm dilated at cesarean section

Exclusion Criteria:

* Patient unwilling or unable to provide informed consent
* Retained placenta or other known cause of postpartum hemorrhage
* Placenta accreta spectrum
* Coagulopathy
* Rupture uterus
* Surgical management immediately needed for life-threatening bleeding
* Known contraindication for Jada System; ongoing intrauterin pregnancy, untreated uterine rupture, unresolved uterine inversion, current cervical cancer, unknown uterine anomoly, current purulent infection

Ages: 18 Years to 44 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Female
Enrollment: 424 (Estimated)
Dates: Start 2023-10-23 (Actual); Primary Completion 2026-08-31 (Estimated); Study Completion 2027-04-30 (Estimated)

PRIMARY OUTCOMES:
Maternal survival without surgical intervention | Delivery to 6 weeks post-delivery
  No maternal death postpartum up to 6 weeks and no use of surgical interventions

SECONDARY OUTCOMES:
Time from randomization to control of bleeding | 6 weeks postpartum
  Time from use of first line treatment to control of bleeding
Concentration of postpartum hemoglobin | Postpartum day 1
  hemoglobin level postpartum
Change in hemoglobin concentration from labor admission to postpartum day 1 | Postpartum day 1
  Hemoglobin change between labor admission and postpartum
Rate of maternal transfusion of blood or blood products postpartum | 6 weeks postpartum
  Transfusion of blood or blood products postpartum
Number of units of blood products transfused | 6 weeks postpartum
  Number of units of blood products transfused
Volume of blood loss post-randomization | 6 weeks postpartum
  An estimate of blood loss from the time of randomization
Surgical procedures performed | 6 weeks postpartum
  Surgical procedures performed, including uterine vascular ligation, uterine compression sutures or hysterectomy
Rate of maternal death postpartum | 6 weeks postpartum
  Maternal death postpartum up to 6 weeks
Number of additional uterotonic used after randomization | 6 weeks postpartum
  Type and number of uterotonic used after the first line oxytocin
Patient satisfaction assessed by a score on a scale of 0 (least satisfied) to 10 (most satisfied) | 6 weeks postpartum
  Patient satisfaction assessed by a score on a scale of 0 (least satisfied) to 10 (most satisfied)
Composite adverse events potentially related to the Jada system | 6 weeks postpartum
  Composite adverse events potentially related to the Jada system, including genital tract injury, uterine perforation or rupture and endometriosis
Quality-adjusted Life-year | 6 weeks postpartum
  Quality-adjusted Life-year based on the literature and Quality of Life Questionnaire (EQ-5D-5L)
Incremental cost per quality-adjusted life-year | 6 weeks postpartum
  Incremental cost per quality-adjusted life-year

CONTACTS AND LOCATIONS:
Overall Officials: Methodius Tuuli, MD, MPH, MBA, Principal Investigator — Women and Infants Hospital of Rhode Island
Locations (2):
- Ghana (2):
  - Komfo Anokye Teaching Hospital, Kumasi, Ashanti Region
  - Korle-bu Teaching Hospital, Accra, Greater Accra Region

IPD SHARING:
Plan to Share IPD: Yes
Data will be collected from human subjects and will be shared according to NIH guidelines. We are committed to the sharing of final data, being mindful that the rights and privacy of people who participate in research must be protected at all times. We will make a complete study dataset available for sharing. We will have a description of study dataset, including code books, meta-data related to the dataset, and documented programming code used for creating the final study population, for creating variables, and for conducting all outcomes analyses. We will remain HIPAA compliant, and therefore any datasets resulting from participants will be free of any identifiers that would permit linkages to individual research participants and variables that could lead to deductive disclosure of individual subjects.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: 5 years after completion of trial.
Access Criteria: We will make the data and associated documentation available to users under a data-sharing agreement that provides for commitment to: a) using the data only for research purposes and not to identify any individual participant; b) securing the data using appropriate computer technology; and c) destroying or returning the data after analyses are completed. Timelines for distribution of data will vary depending on any required restrictions as mentioned above. Data may be distributed by a number of electronic methods, including web-based databases, datasets, and spreadsheets, or via electronic media such as compact discs.